CLINICAL TRIAL: NCT07207109
Title: A Double-blind Randomised Controlled Study to Investigate the Effect of a follow-on Formula With a Specific Synbiotic Mixture on the Gut Microbiota Composition in Healthy Infants.
Brief Title: Effect of follow-on Formula on the Gut Microbiota of Healthy Infants.
Acronym: FUNTASTIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Collaborators: PT Nutricia Indonesia Sejahtera (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 24REX0075490
Record Dates: First submitted 2025-09-23; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Follow-on Formula; Infant; Faeces; Gut Microbiota
Keywords: Follow-on formula; healthy infants; gut microbiota
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test product (Experimental): Group that receives follow-on formula with synbiotics
  Interventions: Other: Test: Follow-on formula with synbiotics
- control product (Active Comparator): Group that receives regular follow-on formula
  Interventions: Other: Control: Regular follow-on formula

INTERVENTIONS:
Other: Test: Follow-on formula with synbiotics — Intervention description: both products are nutritionally complete follow-on formulas
  Arms: test product
Other: Control: Regular follow-on formula — Intervention description: both products are nutritionally complete follow-on formulas
  Arms: control product

SUMMARY:
This study investigates the effects of follow-on formula in infants aged 6-9 months over a 12-week period. After parents give consent, their baby's feeding habits, stool characteristics, and any illnesses or medication use will be recorded. Infants will be randomly assigned to receive either the test or control product. Growth and health data will be collected during study visits.

Parents will collect stool samples and complete diaries to help researchers better understand the baby's digestion and overall health. A follow-up phone call will be made to check on the baby's well-being after the study ends.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants as per the clinical judgement of the Investigator
2. Singleton infants
3. Infants ≥6 months and ≤9 months of age at Visit 1
4. Infant's weight-for-age WHO z-score within ± 2 SD at Visit 1
5. Infants fed with an infant or follow-on formula at Visit 1.
6. Infants are familiar with, and are expected to drink, ≥600 mL formula per day.
7. Written informed consent (IC) from parent(s) and/or legally acceptable representative(s) aged ≥18 years at Visit 1.

Exclusion Criteria:

1. Infants with known or suspected medical conditions requiring a special diet or special formulae, food allergy, or food intolerances
2. Infants who received breastfeeding ≤14 days before Visit 1
3. Infants who are potty-trained
4. Infants with current or previous illnesses/conditions and/or known or suspected congenital diseases or malformations which could interfere with the study outcomes, as per investigator's clinical judgement.
5. Use of medication or nutritional products/food supplements known to impact the study outcomes ≤14 days before Visit 1 or expected need during the study.
6. Infants with previous, current, or intended participation in any other clinical study involving investigational or marketed products.
7. Incapability of infants' parents and/or legally acceptable representative(s) to comply with study protocol as per the judgement of the investigator or investigator's uncertainty about the willingness or ability of parents legally acceptable representative(s) to comply with the protocol requirements, including access to a phone.
8. Children of employees and/or family members or relatives of employees of Danone, the participating sites, or any other nutrition company that develops infant, follow-on or young child formulae.

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 268 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Bifidobacteria proportions | Baseline and 12 weeks postbaseline
  The mean change from baseline in the proportion of faecal Bifidobacterium at 12 weeks postbaseline

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - DPS_RSUP Prof. Dr. I.G.N.G. Ngoerah, Denpasar, Bali
  - SBY_RSUD Dr. Soetomo, Surabaya, East Java

IPD SHARING:
Plan to Share IPD: No